CLINICAL TRIAL: NCT04747106
Title: Thromboelastography Guides a Multicentre Cluster Controlled Study of Plasma Exchange for Hepatitis B Associated Acute on Chronic Liver Failure
Brief Title: Thromboelastography Guides a Multicentre Cluster Controlled Study of Plasma Exchange for Hepatitis B Associated Acute-on-chronic Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Jinjun Chen, Associate Director, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: 28 Day Mortality
MeSH Terms: interventions — Plasma Exchange

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plasma exchange (Experimental): when ADP inhibition >30%, plasma exchange, once or twice a week, 1000-1500ml plasma was exchanged for each time
  Interventions: Biological: plasma exchange
- standard medical treatment (No Intervention): standard medical treatment

INTERVENTIONS:
Biological: plasma exchange — when ADP inhibition >30%, plasma exchange, once or twice a week, 1000-1500ml plasma was exchanged for each time
  Arms: plasma exchange

SUMMARY:
In the past ten years, the extracorporeal liver support system has been widely used in clinical practice as a first-line treatment of liver failure. Plasma exchange (PE) can remove toxic substances in ACLF patients, reduce liver damage, and replenish coagulation factors, albumin and immunoglobulins, thereby improving the liver's microenvironment and accelerating liver regeneration and functional recovery. The ACLF study showed that PE can improve the symptoms of patients and improve the short-term prognosis of patients, but there are still studies showing that PE does not significantly improve the short-term prognosis of patients. Therefore, the therapeutic effect of PE on ACLF is still controversial. We consider that some people may benefit from plasma exchange, and new indicators are needed to guide disease stratification treatment. Our multi-center prospective data show that plasma exchange has a tendency to improve survival in ACLF-2. After stratifying with ADP inhibition rate in ACLF-2, patients with ADP inhibition rate greater than 30% will be treated 28 days after PE treatment. The prognosis is improving. Therefore, we consider that PE is expected to reduce the mortality of patients with ACLF 2 with an ADP suppression rate greater than 30%, but prospective large-sample clinical studies are still needed.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18-80 years old; 2) Chronic HBV infection related: HBsAg positive for more than 6 months; 3) EASL-ACLF grade 2

Exclusion Criteria:

* 1) Other causes of chronic liver disease; 2) Active bleeding and diffuse intravascular coagulation; 3) Those who have been severely allergic to blood products and heparin in the past; 4) Circulatory failure; 5) Respiratory failure; 6) Patients with unstable period of cardiovascular and cerebrovascular infarction; 7) Those who have received platelet transfusion or artificial liver within 1 week; 8) Patients with liver cancer or other malignant tumors; 9) Pregnant and lactating women; 10) Those with other serious chronic diseases; 11) Fail to sign the informed consent form; 12) Circumstances that the researcher considers inappropriate to participate in the research.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No